CLINICAL TRIAL: NCT03618212
Title: MRI in Multiple Myeloma: Analysis of the Axial Skeleton Versus Whole Body. What is the Required Analysis?
Acronym: MYMO
Status: Terminated | Type: Observational
Why Stopped: Departure of the project leader
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOIGCSMERRIL/2016/AL-01
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myeloma patients
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Skeletal MRI and pelvic and spinal MRI

SUMMARY:
The investigators wish to determine which anatomic regions need to be explored in order to correctly diagnose myeloma: whether axial skeletal MRI alone is sufficient or whether it is necessary to perform a total skeletal MRI.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* Patient has been diagnosed with multiple myeloma (> 10% medullary plasma cells + monoclonal protein) or symptomatic myeloma (myeloma + CRAB symptoms (hypercalcemia, renal failure, anemia, bone lesions), or indolent myeloma (myeloma with symptomatic criteria).

Exclusion Criteria:

* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breast feeding
* The patient has an absolute contra-indication for MRI (pace-maker, claustrophobic patient, metal heart valve)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with myeloma as diagnosed according to the International Myeloma Working Group criteria recruited in the service of clinical hematology in either the CHUs of Nîmes or Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Identification of focal lesions ≥ 5mm by axial skeletal MRI of spine and pelvis versus whole-body MRI using diffusion sequences | Day 0
  Fatty tissue replacement by tumoral tissue observed by hyposignal T1 and hypersignal T2 FS or short-TI Inversion Recovery ≥ 5mm

SECONDARY OUTCOMES:
Number of "punched out" lesions ≥ 5mm identified by whole-body MRI with diffusion sequences versus skeletal X-ray | Day 0
Agreement between identification of normal lesions ≥ 5mm by axial skeletal MRI of spine and pelvis versus whole-body MRI using diffusion sequences | Day 0
Agreement between identification of diffuse lesions ≥ 5mm by axial skeletal MRI of spine and pelvis versus whole-body MRI using diffusion sequences | Day 0
Agreement between identification of mixed lesions ≥ 5mm by axial skeletal MRI of spine and pelvis versus whole-body MRI using diffusion sequences | Day 0
Agreement between identification of salt and pepper lesions ≥ 5mm by axial skeletal MRI of spine and pelvis versus whole-body MRI using diffusion sequences | Day 0
Link between type of infiltration and spinal cord karyotype | Day 0
  Yes/no presence of anomaly, and if yes, type of karyotype anomaly
Inter-observer reproducibility for the first 20 patients for the detection of focal lesions ≥ 5mm by axial skeletal MRI of spine and pelvis | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Larbi, MD, Principal Investigator — CHU Nimes
Locations (2):
- France (2):
  - CHU Montpellier, Montpellier
  - CHU Nimes, Nîmes